CLINICAL TRIAL: NCT03554876
Title: Randomized and Controlled Clinical Trial to Evaluate Bacterial Adhesion on Multi-Im® Transepithelial Components Placed on Implants
Brief Title: Randomized and Controlled Clinical Trial to Evaluate Bacterial Adhesion on Multi-Im® Transepithelial Components
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBEA-06-EC/17/Multi-Im
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Biofilm Formation
Keywords: Biofilm; peri-implantitis; metagenomic analysis; abutment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-Im Machined (Active Comparator): Multi-Im Machined
  Interventions: Device: Multi-Im Machined transepithelial component.
- Multi-Im® nanogolden (Experimental): Multi-Im® nanogolden
  Interventions: Device: Multi-Im Nanogolden transepithelial component
- Multi-Im T-Golden (Experimental): Multi-Im T-Golden
  Interventions: Device: Multi-Im Ti-Golden transepithelial component

INTERVENTIONS:
Device: Multi-Im Machined transepithelial component. — Once the implant is placed, the implant loading protocol will be decided following the clinical criteria. When implant loading is to be done, then the Multi-IM machined transepithelial component is connected to the implant.
  Arms: Multi-Im Machined
Device: Multi-Im Nanogolden transepithelial component — Once the implant is placed, the implant loading protocol will be decided following the clinical criteria. When implant loading is to be done, then the Multi-IM Nanogolden transepithelial component is connected to the implant.
  Arms: Multi-Im® nanogolden
Device: Multi-Im Ti-Golden transepithelial component — Once the implant is placed, the implant loading protocol will be decided following the clinical criteria. When implant loading is to be done, then the Multi-IM Ti-Golden transepithelial component is connected to the implant.
  Arms: Multi-Im T-Golden

SUMMARY:
This study evaluates the efficacy of Mutli-Im® transepithelial components in the inhibition of bacterial adhesion.

The control group will be the Multi-Im® transepithelial component with the conventional surface (Multi-IM® Machined) and the experimental group will be the Multi-Im transepithelial components with the Ti-Golden® surface (Multi-Im Golden) or with the nanogolden surface (Multi-Im® nanogolden). Periodontal indices and biofilformation will be assessed during 2 months after implant loading. Metagenomic analysis and PCR technique will be implemented to assess the biofilm formation.

ELIGIBILITY:
Inclusion Criteria:

* Indication of having to place at least three dental implants.
* Plate index ≤ 20% and absence of evidence of active periodontal disease.
* Bleeding index of adjacent teeth ≤ 30%.
* Probing depth in adjacent teeth <4 mm.
* Not having used systemic antibiotics during the last 6 months.
* Non smoker.
* Possibility for observation during the treatment period.
* Having signed the informed consent.

Exclusion Criteria:

* Suffering any alteration or serious hematologic disease.
* Being undergoing or having received in the 30 days prior to inclusion:

radiotherapy, chemotherapy or immunosuppressive treatments, systemic corticosteroids and/or anticoagulants.

* Presence of malignant tumors, hemangiomas or angiomas in the area of implant placement.
* Patients undergoing treatment with bisphosphonate drugs, both orally and intravenously.
* Metabolic bone disease.
* Diseases that affect the oral mucosa.
* Diabetic patients.
* Severe parafunctional habits and/or temporomandibular joint disorders.
* Pregnant or lactating women.
* Physical or mental inability to maintain a good oral hygiene.
* Being participating in another study.
* In general, any inability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Total amount of the 25 most relevant bacterial species in peri-implantitis processes measured in the retired Multi-Im implants | 24 hours
Total amount of the 25 most relevant bacterial species in peri-implantitis processes | 2 months

SECONDARY OUTCOMES:
Total number of bacterial species. | 24 hours, 2 months
Total amount of the 6 most abundant bacterial species. | 24 hours, 2 months
Dental plaque index | Baseline, 24 hours, 2 months
Gingival index of the natural teeth | Baseline, 24 hours, 2 months
Probing depth of natural teeth | Baseline, 24 hours, 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Eduardo Anitua, Vitoria-Gasteiz, Spain

REFERENCES:
- [Derived] Anitua E, Murias-Freijo A, Tierno R, Tejero R, Alkhraisat MH. Assessing peri-implant bacterial community structure: the effect of microbiome sample collection method. BMC Oral Health. 2024 Aug 26;24(1):1001. doi: 10.1186/s12903-024-04675-y. PMID 39187802